CLINICAL TRIAL: NCT05104853
Title: A Phase 2a Double Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Efficacy of CNP-104 in Subjects Ages 18-75 with Primary Biliary Cholangitis Who Are Unresponsive to UDCA And/or OCA
Brief Title: Study to Evaluate the Safety, Tolerability, PDs, and Efficacy of CNP-104 in Subjects with Primary Biliary Cholangitis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: COUR Pharmaceutical Development Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CNP-104-5.001
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4 mg/Kg CNP-104 (Experimental): 200 mL intravenous infusion on Day 1 and Day 8: 4 mg/Kg CNP-104
  Interventions: Drug: CNP-104
- 8 mg/Kg CNP-104 (Experimental): 200 mL intravenous infusion on Day 1 and Day 8: 8 mg/Kg CNP-104
  Interventions: Drug: CNP-104
- Placebo (Placebo Comparator): 200 mL intravenous infusion on Day 1 and Day 8: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNP-104 — CNP-104 is comprised of PDC-E2 peptide dispersed within a negatively charged polymer matrix of poly (lactic-co-glycolic acid) (PLGA) particles at a target concentration of ~1 μg of PDC-E2 peptide per mg of PLGA particles.
  Arms: 4 mg/Kg CNP-104; 8 mg/Kg CNP-104
Drug: Placebo — CNP-104 Placebo
  Arms: Placebo

SUMMARY:
This study is a Phase 2a First-in-Human (FIH) clinical trial to assess the safety, tolerability, pharmacodynamics (PD), and efficacy of multiple ascending doses of CNP-104. The study consists of a 120 day primary study followed by a 20 month long-term safety and durability of response follow-up period.

DETAILED DESCRIPTION:
Subjects ages 18-75 with primary biliary cholangitis will be screened up to 14 days prior to enrollment into the study. Screening will be completed to assess eligibility, obtain vital signs, collect laboratory samples and PD measurements, and to receive a FibroScan for liver fibrosis. Subjects will additionally complete an initial PBC-40 assessment and begin an Itch Diary, a questionnaire and scoring system to be completed by the patient every morning and evening through Day 120 and then monthly through end of study.

Subjects who meet all inclusion and no exclusion criteria after completing the screening visit will be enrolled in the study. Subjects will be randomized on Day 1 in a 1:1 ratio to receive either CNP-104 or Placebo (0.9% Sodium Chloride USP) by intravenous (IV) infusion. Subjects will be administered CNP-104 or Placebo on Day 1 and on Day 8. This study was originally designed with 2 cohorts, Cohort 1 comprised of 6 subjects randomized 1:1 to placebo or 4 mg/kg, and Cohort 2 comprised of up to 34 subjects randomized 1:1 to placebo or 8 mg/kg. Under Protocol Amendment 6 (v7.0), the remaining subjects for Cohort 2 (approximately 16) will be randomized 1:3:1 to placebo, 4 mg/kg, and 8 mg/kg respectively.

Subjects will remain in the clinic on Day 1 and Day 8 from the time of admission (prior to administration of CNP-104 or Placebo) through the final procedure conducted 4 hours post-dose that same day unless an infusion reaction, or other adverse event, requires an extended duration of monitoring. Subjects will be discharged if safety parameters are acceptable to the investigator.

Seven days after the second administration of CNP-104 or Placebo, subjects must return to the clinic for collection of safety labs, PD measurements, and assessment of AEs and medication changes.

Subjects will continue to be followed for 2 years to assess safety, pharmacodynamics, and immunogenicity during the Post-Dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and able to provide Institutional Review Board (IRB) approved written informed consent and privacy language as per national regulations.
2. Men and non-pregnant women, ages 18-75 years inclusive.
3. Subjects with a PBC diagnosis as demonstrated by the presence of 2 or more of the following 3 diagnostic factors:

   1. Alkaline phosphatase > 1.5× ULN for at least 6 months
   2. Positive AMA titer or, if AMA negative or in low titer (<1:40), positive PBC-specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex])
   3. Liver biopsy findings consistent with PBC
4. Subjects who are unresponsive to UDCA and/or OCA after 6 months of treatment at a stable dose as measured by ALP > 1.5× ULN.
5. For subjects on any medication used to treat the symptoms of PBC (ex. UDCA, OCA, seladelpar), subjects must be on a stable dose for a minimum of 3 months prior to enrollment and must agree not to change their dose through study Day 60 unless reviewed by the medical monitor and approved by the site investigator.
6. Subjects with ALP > 1.5× ULN.
7. Subjects with AST and ALT < 5× ULN.
8. Subjects with hemoglobin ≥ 10 g/dL.
9. Subjects with total bilirubin < 2× ULN.
10. Men and women of child-bearing potential (WOCBP) must agree to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, hysterectomy, bilateral tubal ligation, licensed hormonal methods, intrauterine device (IUD) beginning at the time of screening through Day 90.
11. Female subjects who agree not to donate ova starting at initial screening and through Day 90.
12. Male subjects who agree to not donate sperm starting at screening and through Day 90.

Exclusion Criteria:

1. Subjects with a Class B or Class C Child-Pugh score.
2. Subjects with concomitant liver diseases including chronic viral hepatitis B or C, autoimmune hepatitis, PSC, alcoholic liver disease, Wilson's disease, hemochromatosis, or Gilbert's syndrome.
3. Subjects who have previously undergone liver transplantation.
4. Subjects with decompensated liver disease as defined by the presence or history of any of the following:

   * MELD score > 15
   * Hepatic encephalopathy
   * Ascites
   * Hepatorenal syndrome or serum creatinine > 2 mg/dL
   * Total Bilirubin > 3.0 mg/dL
   * INR >1.8 unless on anticoagulation such as Coumadin
   * History of variceal hemorrhage
5. Subjects with a history of cerebrovascular accident in the past 12 months.
6. Subjects with history of myocardial infarction, as defined by any of the following criteria:

   * Development of pathological Q waves with or without symptoms
   * Imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause
   * Pathological findings of a healed or healing myocardial
7. Subjects with chronic kidney disease, as defined by estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 for at least 3 months (per CKD EPI Equation - 2021).
8. Subjects with uncontrolled diabetes, as defined by HbA1c > 7%.
9. Subjects who have used the following medications:

   * Methotrexate within 90 days of screening.
   * Immunotherapy drugs unless approved by the medical monitor.
10. Subjects with a history of tuberculosis or positive PPD skin test.
11. Subjects who have received administration of any live vaccine (other than intranasal Influenza) within 28 days or subunit vaccine within 14 days prior to screening or are planning to receive any vaccination before Day 90.
12. Subjects who have used systemic steroids within 3 months prior to screening.
13. Subjects with laboratory test results at screening or prior to study dosing that are outside the normal limits and considered by the Investigator to be clinically significant.

    Note: This criterion does not apply to liver function tests. Additionally, clinically significant laboratory test results at screening that are related to the condition (PBC) are acceptable as long as all inclusion and no other exclusion criteria are met.
14. Subjects with positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen/antibody as determined at screening.
15. Subjects with a history of or currently active immune disorders other that PBC (including autoimmune disease) unless the condition, after discussion with the Medical Monitor, has been deemed to be acceptable for the subject's participation in this study.
16. Subjects with a history of or current active diseases requiring immunosuppressive drugs (including azathioprine, prednisone, prednisolone, budesonide, cyclosporine, tacrolimus, methotrexate, or mycophenolate mofetil) unless the condition, after discussion with the Medical Monitor, has been deemed to be acceptable for the subject's participation in this study.
17. Subjects with a clinical history of significant cardiovascular disease as determined by the Investigator.
18. Subjects with a complication or medical history of malignancy within past 5 years which, in the Investigator's opinion, makes the subject unsuitable for study participation.
19. Subjects who, in the Investigator's opinion, will be unable to adhere to study procedures.
20. Subjects who have received an investigational therapy other than CNP-104 within 28 days or 5 half-lives, whichever is longer, prior to screening.
21. Subjects with any condition which, in the Investigator's opinion, makes the subject unsuitable for study participation.
22. Known sensitivity to any components of CNP-104.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) | through Study Completion, an average of 720 Days
  Frequency tables will be presented by treatment group for all AEs and SAEs by System Organ Class (SOC) and Preferred Term (PT). Frequency tables will also be produced by treatment group for AEs leading to discontinuation from TP and study, by severity, and by causality. No formal statistical testing will be done
Laboratory safety assessments (hematology, serum chemistry, coagulation panel, urinalysis). | through Study Completion, an average of 720 Days
  Frequency tables of each assessment abnormalities by grade and treatment will be presented. No formal statistical testing will be done.
Serum Cytokines (TNF-α, IL-4, IL-6, IL-10, IL-1β, MCP-1, MIP-1α, IFN-γ) | through CNP-Dosing Period, an average of 15 Days
  Frequency tables will be presented by treatment group. No formal statistical testing will be done

SECONDARY OUTCOMES:
To assess the change from baseline in Serum Alkaline Phosphatase (ALP) levels, for safety only | through Visit 6, an average of 60 Days and Visit 16, an average of 720 Days
  Change from baseline in ALP levels at Day 60 and Day 720
To assess the change from baseline in AMA | through Visit 7, an average of 90 Days and Visit 16, an average of 720 Days
  Change from baseline in AMA between placebo and CNP-104 at Day 90 and Day 720
To assess the change from baseline in liver fibrosis by FibroScan | through Visit 7, an average of 90 Days and Visit 16, an average of 720 Days
  Change from baseline in liver fibrosis by FibroScan between placebo and CNP-104 at Day 90 and Day 720
To assess the change from baseline in modified PBC-40 score | through Visit 6, an average of 60 Days and Visit 16, an average of 720 Days
  Change from baseline in modified PBC-40 score between placebo and CNP-104 at Day 60 and Day 720
To assess the change from baseline in Weekly Mean Itch Score | through Visit 6, an average of 60 Days and Visit 16, an average of 720 D
  Change from baseline in Weekly Mean Itch Score between placebo and CNP-104 at Day 60 and Day 720
To assess the change from baseline in liver enzymes (Albumin, Bilirubin (total and direct), ALT, AST, GGT) | through Visit 6, an average of 60 Days and Visit 16, an average of 720 Days
  Change from baseline in liver enzymes at Days 60 and 720
To assess the change in antigen specific CD4+ and CD8+ T cells | through Visit 6, an average of 60 Days and Visit 16, an average of 720 Days
  Change from baseline in antigen specific CD4+ and CD8+ T at Days 60 and 720

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowlus, MD, Principal Investigator — UC Davis
Locations (19):
- United States (19):
  - Southern California Research Center, Coronado, California
  - OM Research, Lancaster, California
  - University of California Davis Health, Sacramento, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida - Hepatology Research, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - GI PROS Research, Naples, Florida
  - Cleveland Clinic - Florida, Weston, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Texas Liver Institute, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klatzkow H, Bhavsar-Burke I, Pearson M, Wentworth BJ. Primary Biliary Cholangitis in 2025: A New Frontier. Am J Gastroenterol. 2025 Dec 1;120(12):2746-2749. doi: 10.14309/ajg.0000000000003559. Epub 2025 May 29. No abstract available. PMID 40439725